CLINICAL TRIAL: NCT05441397
Title: Prevalence of Periodontitis Based Upon Principles Presented by the 2017 Classification: A Hospital-based Cross-sectional Study on a Sample of Young Egyptian Dental Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Rana Taha Galal El-Hanify, MASTER STUDENT, Cairo University
Other Study IDs: 6322
Record Dates: First submitted 2022-06-28; First posted 2022-07-01 (Actual); Last update posted 2022-07-01 (Actual); Status verified 2022-06

CONDITIONS: Periodontitis
MeSH Terms: conditions — Periodontitis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study aims at determining the Prevalence Of Periodontitis based upon principles presented by the 2017 Classification: A Hospital-Based Cross-Sectional Study on A Sample of Young Egyptian Dental Patients

ELIGIBILITY:
Inclusion Criteria:

1. Patients whose age from 12 to 39 years old .
2. Patient consulting in the outpatient clinic
3. Provide informed consent.

Exclusion Criteria:

1. Patients having problem in opening their mouth or undergoing inter maxillary fixation where oral examination will not be possible.
2. Patients diagnosed with psychiatric problems or intoxicated with alcohol or drugs

Ages: 12 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Young Egyptian dental outpatients attending the oral diagnosis clinic at faculty of Dentistry, Cairo University
Sampling Method: Probability Sample
Enrollment: 464 (Estimated)
Dates: Start 2022-06-30 (Estimated); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-08-30 (Estimated)

PRIMARY OUTCOMES:
Probing pocket depth Staging & Grading | up to 1 day
  UNC-15 periodontal probe
Clinical attachment level | up to 1 day
  UNC-15 periodontal probe

SECONDARY OUTCOMES:
Nutritional status | up to 1 day
  Questionnaire Yes-No

CONTACTS AND LOCATIONS:
Overall Officials: Rana T EL-Hanify, BDs, Principal Investigator — Cairo University; Nesma M Shemais, PHD, Study Director — lecturer of oral medicine and periodontology ,faculty of dentistry ,Cairo university; Weam A el-battawy, PHD, Study Director — associate professor of oral medicine and periodontology ,faculty of dentistry ,Cairo university; Manal M Hosny, PHD, Study Chair — professor of oral medicine and periodontology ,faculty of dentistry ,Cairo university
Locations (1):
- Cairo University, Cairo, Egypt